CLINICAL TRIAL: NCT04588649
Title: The Aging Brain and Cognition: Contribution of Vascular Injury, Amyloid Plaque and Tau Protein to Cognitive Dysfunction After Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 103-7584A
Record Dates: First submitted 2020-09-29; First posted 2020-10-19 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2020-09

CONDITIONS: Post-stroke Dementia; Vascular Mild Cognitive Impairment
MeSH Terms: interventions — THK5351

STUDY DESIGN:
Intervention Model Description: * GroupA (Stroke/TIA patients), n=300
  * Group (healthy elderly controls), n=30
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THK-5351 (Other): Name: [18F]THK5351，(S)-6-[(3-Fluoro-2-hydroxy)propoxy]-2-(2-Methylaminopyrid-5-yl)-quinoline Dosage form: intravenous injection Dose(s): 10mCi Dosing schedule: Visit 2 Mechanism of action (if known): high affinity radiotracer for the tau protein Pharmacological category：Radio pharmaceutical
  Interventions: Drug: THK-5351; Drug: AV-45
- AV-45 (Other): Name: [18F]AV-45, (E)-4-(2-(6-(2-(2-(2-[18F]fluoroethoxy) ethoxy) ethoxy)pyridin-3-yl)vinyl)-N-methylbenzenamine Dosage form: intravenous injection Dose(s): 10mCi Dosing schedule: Visit 2 Mechanism of action (if known): high affinity radiotracer for the β- amyloid protein Pharmacological category：Radio pharmaceutical
  Interventions: Drug: THK-5351; Drug: AV-45

INTERVENTIONS:
Drug: THK-5351 — [18F]THK-5351 PET Imaging
Drug: AV-45 — [18F]AV-45 PET Imaging

SUMMARY:
Stroke can lead to signficiant neurological deficits, and about one-third of stroke patients will be diagnosed of vascular mild cognitive impairment or post-stroke dementia. Post-stroke dementia includes all types of dementia that happen after stroke, irrespective of their cause, and vascular dementia (VaD), degenerative dementia (especially Alzheimer's disease), or mixed dementia (dementia as a result of the coexistence of vascular lesions of the brain and neurodegenerative lesions) are the most common causes of post-stroke dementia. However, it is difficult to determine to what extent cognitive impairment may be attributable to stroke versus concomitant Alzheimer disease. With the advent of PET imaging technique, we are able to conduct a multi-modal neuroimaging study to explore the composite influence of vascular injury, amyloid plaque and Tau protein the the cognitive performance after stroke.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for stroke/TIA patients

* Males or females with age >= 50 years old
* Having cerebral stroke or transient ischemic attack
* Modified Rankin Scale < 4
* Ability to participate in cognitive and neuroimaging assessments
* Female subjects of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception after the final study
* Provision of signed informed consent

Inclusion criteria for healthy elderly controls

* Males or females with age >= 50 years old
* Without history of cerebral stroke or transient ischemic attack
* Ability to participate in cognitive and neuroimaging assessments
* Female subjects of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception after the final study
* Provision of signed informed consent

Exclusion Criteria:

Exclusion criteria for all subjects

* Presence of dementia diagnosis before the index stroke or at the initial screening History of vascular MCI (VaMCI)
* The Chinese version of the Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE) score >=104 [24] at the initial screening.
* Presence of large infarction or lobar encephalomalacia on brain CT or MRI.
* Severe language impairment precluding cognitive assessments, defined as a score of 3 points in the language score of the National Institute of Health Stroke Scale.
* Life expectancy less than 1 year.
* Clinically significant abnormal laboratory values.
* Clinically significant or unstable medical or psychiatric illness.
* Epilepsy history.
* Cognitive impairment resulting from trauma or brain damage.
* Substance abuse or alcoholism in the past 1 year
* General MRI, and / or PET exclusion criteria.
* Pregnant or becoming pregnant during the study (as documented by pregnancy testing at screening or at any date during the study according to the PI discretion) or current breast feeding.
* History of allergy to 18F-labelled radionucleic agents, [18F]AV-45 or [18F]THK-5351.
* Subjects having high risks for the study according to the PI discretion.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2016-03-29 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
CDR score of cognition deteriorating group and stable group | through study completion, an average of 1.5 year
  The CDR is a 5-point scale (0、0.5、1、2、3) used to characterize six domains of cognitive and functional performance applicable to Alzheimer disease and related dementias: Memory, Orientation, Judgment & Problem Solving, Community Affairs, Home & Hobbies, and Personal Care. The necessary information to make each rating is obtained through a semi-structured interview of the patient and a reliable informant or collateral source (e.g., family member).
  Global score 0 = Normal、0.5 = Very Mild Dementia、1 = Mild Dementia、2 = Moderate Dementia、3 = Severe Dementia. The cognition deteriorating group is defined as CDR score declines from 0 or 0.5 at Month 3 to >=1 at Month 18. The cognition stable group is defined as CDR score remains at 0 or 0.5 at Month 18.
Imaging positive and negative conditions | through study completion, an average of 1.5 year
  PET images are visually assessed by independent raters, who are nuclear medicine doctors and blinded to all clinical and diagnostic information. The raters classify each scan as 0-1 (no significant uptake)、2 (suspicious uptake)、3-4 (significant uptake). The score >= 2 is deemed as positive condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, Chang-Gung memorial Hospital, Taoyuan District, Guishan, Taiwan